CLINICAL TRIAL: NCT06343454
Title: Effect of Different Head Positions on Occlusal Contacts
Brief Title: The Effect of Different Head Positions on Occlusal Contacts During Digital Interocclusal Bite Registration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sinem Kahya Karaca, Research Assistant, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2023/04-03(KA-22111)
Record Dates: First submitted 2024-03-22; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Occlusion
Keywords: Occlusal contacts; Head position; Digital occlusal analysis
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neutral Head Position (Other): Neutral head position (PN), in which the head is positioned on the head-neck-spine plane.
  Interventions: Other: Digital Interocclusal Record In Different Head Positions
- Forward Head Position (Other): Forward head position/active feeding position (PF), in which head is positioned 30° in front of head-neck-spine plane with forward head tilt.
  Interventions: Other: Digital Interocclusal Record In Different Head Positions
- Backward Head Position (Other): Backward head position/drinking position (PB), in which the head is positioned 45° behind the head-neck-spine plane with backward head tilt.
  Interventions: Other: Digital Interocclusal Record In Different Head Positions

INTERVENTIONS:
Other: Digital Interocclusal Record In Different Head Positions — Recording the position of the upper and lower teeth in the bite position in different head positions with an intraoral scanner

SUMMARY:
The goal of this clinical trial is to learn about different head position's effect on occlusal contacts during digital interocclusal record. The main question aims to answer is:

• Are different head positions in physiological limits can be affected the occlusal contact during interocclusal record? Participants will be asked to stand in three different physiological head positions (neutral, forward and backward) which are common in daily routine. In these positions, after maxillary and mandibular arch scans three different interocclusal records will be taken. Also for assessment of these records in digital occlusal analysis module (oJMA, zebras), three different oJMA record will be taken.

Researchers will compare neutral, forward and backward head positions to see if there are any difference in number, density and location of occlusal contacts.

DETAILED DESCRIPTION:
The purpose of this clinical study was to compare, within physiological bounds, the occlusal contacts obtained with the interocclusal records taken with an intraoral scanner in three distinct head positions. The clinical protocol was approved by national ethical committees. After the consent form is accepted, those who fit the inclusion criteria will be enrolled in the study. The Power analysis led to the determination that 36 people would be needed to participate in the study.

The possibility of experiencing nausea during surface scanning and interocclusal records is one risk that could arise during the research. But routine scans carry a risk of developing this. It also has nothing to do with the study specifically. The process will end if there is severe nausea, anxiety, restlessness, anxiety during surface scanning, or an oJMA record. Participants will have the option to withdraw from the study at any time before or after enrollment opens. We'll find new people to take their place. Once there is a sufficient number of participants, registrations from these fully dentate individuals who do not require dental treatment will start. Study groups also formed to obtain digital interocclusal records in three head positions: "neutral head position (PN)," in which the head is positioned on the head-neck-spine plane; "forward head position/active feeding position (PF)," in which the head is positioned 30° in front of the head-neck-spine plane with forward head tilt; and "backward head position/drinking position (PB)," in which the head is positioned 45° behind the head-neck-spine plane with backward head tilt. PN considered the control group. The interocclusal records will be taken digitally with an IOS in the mentioned head positions.

Digital recording procedures will start after the examination. The recordings will be completed in two sessions. All recording methods have features that do not damage the oral tissues and do not cause pain or sensitivity. The first session will be completed within 10 minutes. First, a surface scan of the upper and lower jaws will be performed with an intraoral scanner and will be completed within three minutes. All scans will be performed in the entire arch and single-stage, according to the manufacturer's recommendations. Following the scan, missing regions and stitching errors will be monitored, and only scans devoid of these issues will be approved. Direct digital interocclusal records will then be taken and will be repeated for three different head positions. A manual goniometer (Goniometer, 360°; Saehan, Germany) will be used to determine the head position. The patient's head will next be adjusted to the predetermined position by using the dental chair's head support, and a goniometer will be used to confirm the adjustment. The interocclusal record will be performed in a static position, keeping the head fixed in the specified position. The record will be completed by starting from the most posterior tooth possible, moving horizontally anteriorly, and then posteriorly in the same direction. The same process will be repeated for the left interocclusal record. All interocclusal records will be achieved with auto-alignment.

The "digital occlusion analysis module" in the WINJAW+RC software program of oJMA will be used for detailed analysis of occlusal contacts. In the second session, the interocclusal records taken in the PN position will be transferred to this analysis module, and the necessary oJMA records will be. Before the oJMA record, the patient will be seated in the dental unit so that the head-neck-spine plane is perpendicular to the floor and the dental unit supports the back and head. Three oJMA recordings for the digital occlusion analysis module (oJMA, zebris) will be made, and these recordings will be used to assess the contacts that were previously acquired using the interocclusal records. The maxilla's three-dimensional (3D) position relative to the skull base and the lower jaw position record required for the digital occlusion module will be recorded. The evaluation will be performed by a single investigator using the digital occlusion analysis module, comparing the number, density, and location of occlusal contacts of the posterior teeth in the right and left quadrants in three different head positions. Within this area, cross-sections will be taken at 1mm intervals in the bucco-lingual (BL) direction with fixed x, y, and z coordinates. In each subject, the number of evaluated consecutive cross-sections in each quadrant will be determined. Each cross-section will be evaluated for the presence or absence of a contact point, the number and shape of the contact (point or area), the contact point's density, and the contact's anatomical location on the occlusal surface of the tooth. Each contact assessment will be expressed qualitatively as either present (1) or absent (0). A value of "1" will be given for each contact and all conditions obtained for its characteristics, and these values will be summed. This number will be divided by the total number of sections evaluated. Data will be generated based on this proportional value.

The comparison and statistical evaluation of these data with computer software constitute the experimental part of this study. The qualitative variables of all patients included in this study will be described with numbers and percentages. IBM SPSS Statistics 25 will be used for the data analysis. The Kolmogorov-Smirnov normality test will assess the data's conformity to a normal distribution. The Paired Samples t-test will be used to compare the data groups that are determined to be suitable for a normal distribution. The statistical significance level will be set at 0.05.

Each patient will be named by numbers (1, 2, 3...) and head position codes (PN, PB, PF), and no individual data will be included. Personal data will not be included in any software to be used during the study, will not be shared with anyone, and will remain confidential only with the physician. The surface scans and recording process will not provide any direct benefit for the participants. The results of this study can be used in dental education or scientific publications without revealing the patient's identity.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 18 years of age,
* Individuals with natural dentition,
* Individuals with healthy head and neck movements within physiologic limits, - Individuals with Angle Class I skeletal relation
* Individuals with stable maximum intercuspal relation and absence of premature tooth contact.
* Individuals with radiologic and periodontal health of the teeth.

Exclusion Criteria:

* Individuals with general health problems
* Individuals with missing teeth
* Individuals with lack of posterior occlusal support or unstable occlusion
* Individuals with pain in the orofacial region and TMJ disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-01-27 (Actual); Study Completion 2024-03-03 (Actual)

PRIMARY OUTCOMES:
Number of Occlusal Contacts | Up to 24 weeks
  Evaluating the number of contacts in terms of point and area contact.
Density of Occlusal Contacts | Up to 24 weeks
  Evaluating the contact density by dividing the density in three groups (low, medium, and high).
Location of Occlusal Contacts | Up to 24 weeks
  Evaluating the location of contacts in "functional cusp," "central fossa," and "non-functional cusp." sections.

CONTACTS AND LOCATIONS:
Overall Officials: Sinem Kahya Karaca, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haralur S, Al-Gadhaan S, Al-Qahtani A, Mossa A, Al-Shehri W, Addas M. Influence of functional head postures on the dynamic functional occlusal parameters. Ann Med Health Sci Res. 2014 Jul;4(4):562-6. doi: 10.4103/2141-9248.139319. PMID 25221705
- [Background] Gupta S, Tarannum F, Gupta NK, Upadhyay M, Abdullah A. Effect of head posture on tooth contacts in dentate and complete denture wearers using computerized occlusal analysis system. J Indian Prosthodont Soc. 2017 Jul-Sep;17(3):250-254. doi: 10.4103/jips.jips_321_16. PMID 28936038
- [Result] Chapman RJ, Maness WL, Osorio J. Occlusal contact variation with changes in head position. Int J Prosthodont. 1991 Jul-Aug;4(4):377-81. PMID 1811633
- [Result] Kordass B, Amlang A, Hugger A, Behrendt C, Ruge S. Number and localization of occlusal contact areas on natural posterior teeth without dental findings - evaluations of the regional baseline study (SHIP-1) with the Greifswald Digital Analyzing System (GEDAS). Int J Comput Dent. 2022 Mar 24;25(1):47-56. PMID 35322652

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT06343454/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT06343454/ICF_001.pdf